CLINICAL TRIAL: NCT00831402
Title: Assessment of Thyroid Function Throughout Pregnancy With and Without Iodine Supplementation
Brief Title: Thyroid Function Throughout Pregnancy With and Without Iodine Supplementation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 05-PHRC-03
Record Dates: First submitted 2009-01-28; First posted 2009-01-29 (Estimated); Last update posted 2024-03-18 (Actual); Status verified 2009-02

CONDITIONS: Pregnancy
Keywords: woman

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm without iodized vitamin (VITAMIN OLIGOBS PREGNANCY) (Other): 50 women will be studied in the absence of iodized supplémentation(natural history of function thyroïdienne in the course of the pregnancy and in the post partum)
  Interventions: Dietary Supplement: controll group
- Arm with iodized vitamin (Active Comparator): The 50 women will be follow up with a supplémentation iodized by vitamins of pregnancy strengthened in iodin everything in the course of the pregnancy and during the 3 months post partum (Oligobs Maxiode, 150 mcg / of iodizes, is 2cp a day)
  Interventions: Dietary Supplement: Oligobs Maxiode

INTERVENTIONS:
Dietary Supplement: Oligobs Maxiode — The 50 women will be follow up with a supplémentation iodized by vitamins of pregnancy strengthened in iodin everything in the course of the pregnancy and during the 3 months post partum (Oligobs Maxiode, 150 mcg / of iodizes, is 2cp a day)
  Arms: Arm with iodized vitamin
Dietary Supplement: controll group — 50 women will be studied in the absence of iodized supplémentation(natural history of function thyroïdienne in the course of the pregnancy and in the post partum)
  Arms: Arm without iodized vitamin (VITAMIN OLIGOBS PREGNANCY)

SUMMARY:
Goals of the study :

1. To study maternal thyroid function during pregnancy with or without supplementation with pregnancy tablets fortified with iodine
2. To establish reference values of thyroid function at different stages of pregnancy (3 trimesters)
3. To precise screening strategy of iodine deficiency in our population and suggest recommendation for its prevention.

DETAILED DESCRIPTION:
Overt maternal hypothyroidism and/or iodine deficiency during pregnancy are linked to mental retardation in their offspring. Iodine deficiency may lead to maternal hypothyroxinemia, and even mild hypothyroidism in predisposed women. Indeed, thyroid hormones are of paramount importance for fetal brain development. During the first trimester of pregnancy, the only thyroid hormones available to the fetus are from maternal origin. Later in pregnancy, fetal thyroid progressively starts producing thyroid hormone, providing that maternal iodine status is adequate (≥200-250 mcg/day). It has been shown recently that mild maternal hypothyroidism may be responsible for discrete neuropsychological impairment in her child, implying a potential benefit for early screening and care during pregnancy. Furthermore, iodine deficiency is extremely common in our area (Brucker-Davis et al 2004). However, there is no official recommendation for screening and prevention, as for gestational diabetes for example.

We propose to study healthy pregnant women, screened before 12 weeks of gestation and without thyroid disease. They will be randomized in 2 groups and will therefore take pregnancy tablets, iodine fortified or not (Oligobs Maxiode -150 mcg/j of iodine, vs Oligobs grossesse), in addition to appropriate nutritional advice. Their longitudinal study will involve:

1. Evolution of thyroid function parameters in the 2 groups, with comparison of maternal thyroid volumes, maternal thyroid hormones levels and cord blood parameters, including thyroglobulin, during pregnancy and in postpartum.
2. Establishment of reference ranges for thyroid parameters for each trimester of pregnancy.

This public health project rests on our expertise in the care of pregnancies with maternal endocrine and metabolic disease (Hieronimus et al 2003-2005) and on a close collaboration of our Departments within the Pole "Mother-Child", conveniently located at the same hospital. It will allow us to precise iodine deficiency screening and prevention in our population and to structure and optimize the care for women with thyroid disease screened early in pregnancy (opening of a specific clinic), in order to improve maternal and fetal prognosis

ELIGIBILITY:
Inclusion Criteria:

* All women follow-up in the three months of the pregnancy in the CHU de Nice
* Maternal thyroid function is between and 0.1<TSH<2.5 mUI/l, 23>T4L>12 pmol/l
* Person over 18
* Signed lit Consent
* Give birth in the CHU of Nice

Exclusion Criteria:

* Allergy known in iodine
* Iodized surcharge defined by an iodurie> 400 mcg / l
* Catch of ongoing iodized vitamins of pregnancy
* Participation in another research protocol

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 111 (Actual)
Dates: Start 2007-06; Primary Completion 2007-07 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
• Intra individual variation of maternal thyroglobulin between the first trimester and the delivery • And cord blood thyroglobulin With comparison of the 2 groups (control and supplementation with iodine) | Every 3 months up to the give birth, the day of a give birth, and after three months

SECONDARY OUTCOMES:
Comparison of control and treated groups for : • Frequence of miscarriage, duration of gestation, birth weight, APGAR, neonatal complications, Maternal thyroid function, Frequency of post partum thyroiditis,Cord blood thyroid function | Every 3 months up to the give birth, the day of a give birth, and after three months

CONTACTS AND LOCATIONS:
Overall Officials: Françoise Dr BRUCKER-DAVIS, PH, Principal Investigator — CHU de Nice - Service d'endocrinologie - Hôpital de l'Archet - 151 Route de saint-antoine de ginestière 06200 Nice
Locations (1):
- CHU de Nice - 4 avenue Reine Victoria - Hôpital de Cimiez, Nice, Alpes-Maritimes, France